CLINICAL TRIAL: NCT04587635
Title: Evaluation of Changes in Bowel Movement Frequency Following the Consumption of Partially Hydrolyzed Guar Gum (PHGG) in Adults with Constipation
Brief Title: Evaluation of Changes in Bowel Movement Frequency Following the Consumption of PHGG in Adults with Constipation
Acronym: TYPHOON
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 19.19.CLI
Record Dates: First submitted 2020-09-24; First posted 2020-10-14 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Constipation - Functional

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double blind study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PHGG fiber (Active Comparator): PHGG Fiber
  Interventions: Dietary Supplement: PHGG
- Placebo Maltodextrin (Placebo Comparator): Maltodextrin
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: PHGG — PHGG
  Arms: PHGG fiber
Dietary Supplement: Placebo — Maltodextrin
  Arms: Placebo Maltodextrin

SUMMARY:
Evaluation of Changes in Bowel Movement Frequency Following the Consumption of Partially Hydrolyzed Guar Gum (PHGG) in Adults with Constipation

ELIGIBILITY:
Inclusion criteria:

1. Men or women aged 18-75, inclusive.
2. Self-reported symptoms of constipation for a minimum of 3 months.
3. Constipation symptoms according to the adapted Rome IV Diagnostic Questionnaire for Adults for Functional Constipation (Appendix 2) administered at screening.
4. Cleveland Clinic constipation score (CCCS) of 8-20.
5. Low-moderate fiber intake (≤18g) determined by the semi-quantitative food intake screener known as the Block Fiber Screener completed by site personnel.
6. Ability to understand the participant information sheet and instructions, and able to provide informed consent.
7. Access to a suitable smartphone device (Android or iOS) with ability to download and complete the study e-Diary daily for the duration of the trial.

Exclusion criteria:

1. Pregnant women or breastfeeding.
2. Ongoing other diagnosed gastrointestinal disease or complication (Crohn's disease, Ulcerative Colitis, Coeliac disease, chronic diarrhoea).
3. Any clinically relevant abnormalities in the screening visit physical examination or alarm features in the medical history such as sudden unintentional weight loss (>10% in 3 months), frequent rectal bleeding not caused by anal fissures or hemorrhoids, recent change in bowel habit (<3 months), severe abdominal pain and stool positive for occult blood.
4. Prior abdominal surgery (including gastric bypass or laparoscopic banding), except cholecystectomy and appendectomy.
5. Neurologic diseases such as multiple sclerosis, stroke, spinal cord injury, Hirschsprung disease.
6. Chronic usage of any medication that in the opinion of the investigator would impact gut motility two weeks prior to the initial administration of study product or up to a minimum of 5 times the half-life of the medication if it has a long half-life.
7. Illness that may preclude the participant's ability to complete the study or that may confound the study outcomes (e.g. bowel cancer, prostate cancer, terminal illness, severe cardiovascular disease, chronic renal failure or eating disorders) or any other serious illness resulting in >2 weeks inability to work in the 3 months before the study start.
8. Participants with co-morbid illnesses such as cardiovascular, endocrine, renal or other chronic disease likely to affect gut motility or limit normal functions (e.g. reduced mobility or increased fragility).
9. Ongoing alcohol, drug, or medication abuse (anamnesis only).
10. Self-reported symptoms of pelvic organ prolapse, such as feeling of pressure or fullness in the pelvic area, intra vaginal discomfort, painful intercourse and urinary problems.
11. Moderate or severe active local anorectal problems such as recurrent anal fissures, frequent bleeding, large prolapsing haemorrhoids.
12. Regular use of fiber (e.g. Fybogel, Lactulose) (i.e. no more than 1 standard dose) over the week prior to the screening visit and no more than 6 standard doses in the past 1 month prior to the screening visit.
13. Consumption of any type of yoghurts or probiotic-containing products, i.e. any commercially available product specified as containing Lactobacillus, Bifidobacteria, Streptococcus, Saccharomyces such as Activia, Actimel, Yakult, in the 4 weeks prior to randomization (V0).
14. Participation in another study with any investigational product within 6 months of screening.
15. Participation in another constipation trial in the past year.
16. Investigator believes that the participant is physically or mentally unfit to participate in the trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2020-09-16 (Actual); Primary Completion 2021-11-05 (Actual); Study Completion 2021-11-05 (Actual)

PRIMARY OUTCOMES:
SBM | Baseline to end of treatment, up to 6 weeks.
  Change in mean frequency of Spontaneous Bowel Movements (SBM) as measured by the daily bowel diary from baseline to Week 6 in the treatment group compared to placebo. Frequency will be defined as the mean number of SBM for the 2-week run-in period prior to V0 and the final 2-week period of the intervention period.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Muckley, FRCPI, Principal Investigator — Altantia Food Clinical Trial
Locations (1):
- Atlantia Food Clinical Trial, Cork, Ireland

IPD SHARING:
Plan to Share IPD: No